CLINICAL TRIAL: NCT04456595
Title: Double-Blind, Randomized, Placebo-Controlled Phase III Clinical Trial to Evaluate Efficacy and Safety in Healthcare Professionals of the Adsorbed COVID-19 (Inactivated) Vaccine Manufactured by Sinovac
Brief Title: Clinical Trial of Efficacy and Safety of Sinovac's Adsorbed COVID-19 (Inactivated) Vaccine in Healthcare Professionals
Acronym: PROFISCOV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Collaborators: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COV-02-IB
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Vaccines; sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adult - Vaccine (Experimental): Participants aging 18-59 years receiving two doses with 14-days interval of Adsorbed COVID-19 (inactivated) Vaccine
  Interventions: Biological: Adsorbed COVID-19 (inactivated) Vaccine
- Elderly - Vaccine (Experimental): Participants aging 60 years or above receiving two doses with 14-days interval of Adsorbed COVID-19 (inactivated) Vaccine
  Interventions: Biological: Adsorbed COVID-19 (inactivated) Vaccine
- Adult - Placebo (Placebo Comparator): Participants aging 18-59 years receiving two doses with 14-days interval of placebo
  Interventions: Biological: Placebo
- Elderly - Placebo (Placebo Comparator): Participants aging 60 years or above receiving two doses with 14-days interval of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Adsorbed COVID-19 (inactivated) Vaccine — Adsorbed COVID-19 (inactivated) Vaccine manufactured by Sinovac
  Other Names: CoronaVac
  Arms: Adult - Vaccine; Elderly - Vaccine
Biological: Placebo — Placebo of Adsorbed COVID-19 (inactivated) Vaccine manufactured by Sinovac
  Arms: Adult - Placebo; Elderly - Placebo

SUMMARY:
This is a phase III clinical trial to assess efficacy and safety of the Adsorbed COVID-19 (inactivated) vaccine manufactured by Sinovac in health care professionals

DETAILED DESCRIPTION:
This is a phase III clinical trial to assess efficacy and safety of the Adsorbed COVID-19 (inactivated) vaccine manufactured by Sinovac in health care professionals.

The study will be double-blind placebo-controlled trial with participants randomly allocated 1:1 to placebo and vaccine arms.

The immunization schedule is two doses intramuscular injections (deltoid) with a 14-days interval.

For efficacy, the study aims to detect COVID-19 cases, defined as symptomatic SARS-CoV-2 infections, after the second week post-immunization schedule.

For safety and immunogenicity, participants are categorized in two age groups, Adults (18-59 years) and Elderly (60 years and above). Safety database aims to detect adverse reactions with frequency of 1:1000 or higher in adults and 1:500 in elderly.

All participants will be followed up to 12 months. Interim preliminary efficacy analysis can be triggered by reaching the target number of 61 cases. Primary efficacy analysis requires 151 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years of age or older;
2. Healthcare professionals who work in direct contact care of people with possible or confirmed COVID-19 cases;
3. Agree with periodic contacts by phone or electronic means, and home visits;
4. Show voluntary intention to participate in the study, documented by the informed consent form signed by participant.

Exclusion Criteria:

1. For females: Pregnancy (confirmed by positive beta-hCG test), breastfeeding or intent to engage in sexual relations with reproductive intent without use of birth control methods in the three months following vaccination;
2. Evidence of uncontrolled neurological, cardiac, pulmonary, hepatic or renal disease, according to anamnesis or physical examination. Significant changes in treatment or hospitalizations due to worsening of the condition in the last three months are indicators of uncontrolled disease;
3. Diseases with impaired immune system including: neoplasms (except basal cell carcinoma), congenital or acquired immunodeficiencies and autoimmune diseases not controlled according to anamnesis or physical examination. Significant changes in treatment or hospitalizations due to worsening of the condition in the last three months are indicators of uncontrolled disease;
4. Behavioral, cognitive or psychiatric disease that, in the opinion of the principal investigator or his or her representative physician, affects the participant's ability to understand and cooperate with all study protocol requirements;
5. Any alcohol or drug abuse over the 12 months prior to enrollment in the study that has caused medical, professional or family problems, indicated by clinical history;
6. History of severe allergic reactions or anaphylaxis to the study vaccine or to components thereof;
7. History of asplenia;
8. Participation in another clinical trial with an investigational product in the six months prior to enrollment in the study or planned participation in another clinical trial within the two years following enrollment;
9. Previous participation in a study to evaluate a COVID-19 vaccine or prior exposure to a COVID-19 vaccine;
10. Use of immunosuppressant therapy regimens within the six months prior to enrollment in the study for planned use within the two years following enrollment. Immunosuppressant therapy regimens include: antineoplastic chemotherapy, radiation therapy and immunosuppressants to induce transplant tolerance, among others.
11. Use of immunosuppressive doses of corticosteroids within the three months prior to the enrollment in the study and planned use of immunosuppressive doses of corticoids within the three months following enrollment in the study. Immunosuppressive doses of corticosteroids will be considered the equivalent prednisone 20 mg/day for adults, for longer than one week. Continued use of topical or nasal corticosteroids is not considered an immunosuppressant;
12. Received blood products (transfusions or immunoglobulins) within the three months prior to enrollment in the study, or planned administration of blood products or immunoglobulins within the two years following enrollment in the study;
13. Suspected or confirmed fever within the 72 hours prior to vaccination or axillary temperature greater than 37.8 °C* on the day of vaccination (enrollment may be postponed until participant has gone 72 hours without fever);
14. Possible or confirmed case of COVID-19 on the day of vaccination (vaccination can be postponed until the participant completes 72 hours without symptoms or the diagnosis is ruled out);
15. Received live attenuated virus vaccine or inactivated vaccine within the 28 days or 14 days, respectively, prior to enrollment in the study, or immunization planned within the 28 days after enrollment in the study;
16. History of bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture
17. Any other condition that, in the opinion of the principal investigator or his/her representative physician, could put the safety/rights of potential participants at risk or prevent them from complying with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12688 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Incidence of COVID-19 cases after two-doses immunization schedule | Two weeks after second dose up to one year after first dose
  Number of virologically-confirmed symptomatic COVID-19 two weeks after second dose of vaccine
Frequency of adverse events up to seven days after immunization | Seven days after each immunization
  Frequency of adverse reaction in the seven days following each immunization per age group

SECONDARY OUTCOMES:
Incidence of COVID-19 cases after two-doses immunization schedule according to previous exposure | Two weeks after first dose up to one year after first dose
  Number of virologically-confirmed symptomatic COVID-19 two weeks after second dose of vaccine according to previous exposure to SARS-CoV-2
Incidence of COVID-19 cases after 14-days of first immunization | Two weeks after last dose uup to one year after first dose
  Number of virologically-confirmed symptomatic COVID-19 two weeks after first dose of vaccine, regardless the vaccination schedule was completed
Combined incidence of SARS-CoV-2 infection | Two weeks after second dose up to one year after first dose
  Number of virologically-confirmed and or serologically-confirmed SARS-CoV-2 infections two weeks after first dose of vaccine
Incidence of severe COVID-19 cases after two-doses immunization schedule | Two weeks after second dose up to one year after first dose
  Number of virologically-confirmed severe COVID-19 two weeks after second dose of vaccine
Frequency of adverse events up to 28 days after immunization | 28 days after each immunization
  Frequency of adverse reaction in the 28 days following each immunization per age group
Frequency of severe COVID-19 cases | From first vaccination up to one year after first dose
  Frequency of virologically-confirmed severe COVID-19 cases after receiving, at least, one dose of the vaccine
Frequency of adverse events of special interest after immunization | From first vaccination up to one year after first dose
  Frequency of adverse events of special interest after receiving, at least, one dose of the vaccine
Seroconversion rate | Two weeks after each vaccination
  Number of seroconversion responses to SARS-CoV-2 in the second week after each vaccination per age group in a subset of participants
Cell-mediated immune profile | Two and four weeks afer each vaccination
  Number of cell-mediated immune response against SARS-CoV-2 in the week two and four after the second vaccination per age group in a subset of participants
Seropositivity rate | Two weeks after second vaccination
  Number of seropositive responses to SARS-CoV-2 in the second week after each vaccination per age group in a subset of participants

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Palacios, MD, PhD, Study Director — Butantan Institute
Locations (16):
- Brazil (16):
  - Universidade de Brasília, Brasília, Federal District
  - Hospital Universitário Maria Aparecida Pedrossian, Campo Grande, Mato Grosso do Sul
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Universitário Júlio Müller, Cuiabá, Mount
  - Hospital das Clínicas da Universidade Federal do Paraná, Curitiba, Paraná
  - Hospital Escola da Universidade Federal de Pelotas, Pelotas, Rio Grande do Sul
  - Hospital São Lucas da Pontificia Universidade Catolica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor - Fundação Pio XII, Barretos, São Paulo
  - Hospital das Clínicas da UNICAMP, Campinas, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Universidade Municipal de São Caetano do Sul, São Caetano do Sul, São Paulo
  - Faculdade de Medicina de São José do Rio Preto - FAMERP, São José do Rio Preto, São Paulo
  - Instituto de Infectologia Emílio Ribas, São Paulo, São Paulo
  - Centro de Pesquisas Clínicas do Instituto Central do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo
  - Instituto Israelita de Ensino e Pesquisa Albert Einstein, São Paulo, São Paulo
  - Instituto de Infectologia Evandro Chagas - Fiocruz, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palacios R, Patino EG, de Oliveira Piorelli R, Conde MTRP, Batista AP, Zeng G, Xin Q, Kallas EG, Flores J, Ockenhouse CF, Gast C. Double-Blind, Randomized, Placebo-Controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of treating Healthcare Professionals with the Adsorbed COVID-19 (Inactivated) Vaccine Manufactured by Sinovac - PROFISCOV: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Oct 15;21(1):853. doi: 10.1186/s13063-020-04775-4. PMID 33059771
- [Derived] Luan N, Li T, Wang Y, Cao H, Yin X, Lin K, Liu C. Th2-Oriented Immune Serum After SARS-CoV-2 Vaccination Does Not Enhance Infection In Vitro. Front Immunol. 2022 Apr 8;13:882856. doi: 10.3389/fimmu.2022.882856. eCollection 2022. PMID 35464483